CLINICAL TRIAL: NCT01909323
Title: Digestive Tolerance and Postprandial Glycaemic and Insulinaemic Responses Evaluation of Different Maltitol/FOS Mixtures in Healthy Adults
Brief Title: Digestive Tolerance of Maltitol and FOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syral (Industry)
Collaborators: Beghin-Meiji (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SMALTO
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Digestive Tolerance in Healthy Adults
MeSH Terms: interventions — maltitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- sugary dessert cream (Placebo Comparator)
  Interventions: Other: Placebo
- maltitol alone (Experimental)
  Interventions: Other: maltitol alone
- maltitol 85% / FOS 15% (Experimental)
  Interventions: Other: maltitol 85% / FOS15%
- maltitol 68% / FOS 32% (Experimental)
  Interventions: Other: maltitol 68% / FOS 32%
- maltitol 50% / FOS 50% (Experimental)
  Interventions: Other: maltitol 50% / FOS 50%
- FOS alone (Experimental)
  Interventions: Other: FOS alone

INTERVENTIONS:
Other: maltitol 85% / FOS15%
  Arms: maltitol 85% / FOS 15%
Other: maltitol alone
  Arms: maltitol alone
Other: maltitol 68% / FOS 32%
  Arms: maltitol 68% / FOS 32%
Other: maltitol 50% / FOS 50%
  Arms: maltitol 50% / FOS 50%
Other: FOS alone
  Arms: FOS alone
Other: Placebo
  Arms: sugary dessert cream

SUMMARY:
Digestive symptoms following consumption of low digestibe carbohydrates are generally assessed product by product but several ingredients can be used simultaneously. The study aimed at evaluating to digestive tolerance of maltitol and FOS used in a same food.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30
* normal and regular stool frequency: at least 3 stools per week and no more than 3 per days
* subjects not sufferinf from a metabolic, functional or inflammatory disease affecting intestinal transit and nutrients absorption
* subjects not sufferinf from IBS according to Rome III criteria
* subjects not using mdeiction which could affect nutrients absoprtion

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Composite score of gastrointestinal symptoms in the 24h following the consumption of products | 24 hours

SECONDARY OUTCOMES:
Individual scores of gastrointestinal symptoms: bloating, abdominal discomfort, borborygms, flatulences | 24 and 48 hours
Stool frequcency and consistency | 24 & 48 hours
Glycaemic response | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Gendre, MD, Principal Investigator — Biofortis SAS
Locations (1):
- Biofortis SAS, Saint-Herblain, France